CLINICAL TRIAL: NCT05423847
Title: Point-of-care Ultrasound for the Diagnosis and Risk Stratification of Lower Respiratory Tract Infections in TB Endemic Regions: a Multicenter Prospective Cohort Study
Brief Title: Triage UltraSound in Tb Endemic Regions
Acronym: TrUST
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: National University Hospital for tuberculosis, Cotonou, Benin (Unknown); Ecole Polytechnique Fédérale de Lausanne (Other); University of Witwatersrand, South Africa (Other); National University Hospital (CNHU point G), Bamako, Mali (Unknown)
Responsible Party: Principal Investigator, Dr Boillat-Blanco Noemie, Principal investigator, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CGRB11362
Record Dates: First submitted 2022-03-20; First posted 2022-06-21 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2023-08

CONDITIONS: Tuberculosis; Lower Resp Tract Infection; Pneumonia
MeSH Terms: conditions — Tuberculosis; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood Plasma Urine Nasopharyngeal swab Oropharyngeal swab Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Benin1: Benin urban recruitment site National teaching hospital for tuberculosis, outpatient emergency department
  Interventions: Diagnostic Test: POCUS
- Mali1: Mali urban recruitment site University Hospital Bamako, outpatient emergency department
  Interventions: Diagnostic Test: POCUS
- South-Africa1: South-Africa rural recruitment site 1 Tintswalo hospital, outpatient emergency department
  Interventions: Diagnostic Test: POCUS
- South-Africa2: South-Africa rural recruitment site 2 Zithulele hospital, outpatient emergency department
  Interventions: Diagnostic Test: POCUS

INTERVENTIONS:
Diagnostic Test: POCUS — POCUS of lungs, pericardium and abdomen

SUMMARY:
In Sub-Saharan Africa, lower respiratory tract infections (LRTIs) and tuberculosis (TB) jointly are the leading cause of overall mortality. There is a need to integrate sustainable triage and management strategies into standard care. The TrUST study investigates the utility of point-of-care ultrasound (POCUS) for diagnosis and prognosis of LRTIs in TB endemic regions in the outpatient triage setting. Automated interpretation of POCUS by artificial intelligence (AI) may further standardize and improve its predictive utility as well as facilitate its implementation into usual practice.

DETAILED DESCRIPTION:
Design International multicentre prospective cohort study

Setting This study aims to explore the performance of POCUS in a pre-hospital setting in countries with different prevalences of HIV: South- Africa (high prevalence), Benin (low prevalence) and Mali (low prevalence).

Study procedures Pre-recruitment training Before initiating the study, participating clinicians will benefit from lung ultrasound (LUS) and POCUS protocols for extra pulmonary TB (FASH+ exam) training with a field expert. The participating clinicians are required to pass a final expert test before start of patient recruitment and to have a minimum of 20 supervised US.

Inclusion (Day 0) Patients inclusion will be performed over a period of 18 to maximum 24 months. Recruitment will stop before the anticipated end if the inclusion of 1000 patients is reached.

Clinical data Data collected include demographic characteristics (age, sex, occupation etc.), past medical history (previous TB, Coronavirus Disease (COVID), vaccination status, documented past episodes of COVID-19, HIV status,…), symptoms (respiratory symptoms, specific COVID-19 symptoms (from the Centers for Disease Control COVID checklist), specific pulmonary TB symptoms (from the CDC TB checklist) and routine clinical examination findings (vital parameters, oxygen saturation, lung auscultation,…).

Laboratory analyses

Analyses performed on site:

* HIV screening with a serial two rapid test algorithm as per World Health Organization (WHO) guidelines : Screening with Alere Determine combo®; if positive, confirmation by a second rapid test First Response® HIV 1-2-0, CD4 count and/or Viral load as per national guidelines.
* Sputum for GeneXpert Mycobacterium Tuberculosis (MTB)/rifampicine (RIF) assay
* Induced sputum for a new GeneXpert MTB assay if a routine spot and second morning GeneXpert MTB is negative and sputum quality was low (salivary) as per WHO consolidated guidelines
* Sputum for Gram stain and standard bacteriological culture
* Nasopharyngeal swab for Severe Acute Respiratory Syndrome Coronovirus (SARS-CoV-2) real-time polymerase chain reaction (RT-PCR) (Cepheid Xpert Xpress SARS-CoV-2) Since the additional diagnostic yield of mycobacterial culture is shown to be very low in adult patients with cough in Benin, it is reserved for GenXpert MTB/RIF resistant cases, specimens other than sputum (e.g. pleural effusions, where sensitivity of GeneXpert MTB/RIF is low) and patients with treatment failure. Mycobacterial culture will be done on solid medium (Löwenstein-Jensen).

Analyses performed retrospectively on stored samples:

* Nasopharyngeal swab: PCR for influenza
* Sputum: syndromic molecular panel targeting influenza and atypical bacteria. Radiological examinations
* Chest X-Ray (CXR) - face: digital format will be stored
* LUS exam using a standard point-of-care ultrasound device (ultrasound-on-a-chip), LUS will be recorded according to a standard 12-point acquisition protocol with 4 additional apical sites (2 subclavicular and 2 axillary) for improved TB detection.
* This involves scanning both apexes, the anterior and posterior apexes, anterior superior, anterior inferior, posterior superior, posterior inferior and lateral thorax regions
* FASH plus exam using a standard point-of-care ultrasound device. The FASH plus protocol will be performed in a standardized manner as previously described.

All US images captured will be digitally recorded and transferred via a secured internet connection along with relevant metadata to a secure server for storage. For study quality control purposes, the quality of the image and the interpretation of a random sample of images will be evaluated retrospectively by an experienced radiologist.

Clinician-evaluated LUS and FASH All LUS and FASH exams will be read by 2 independent readers blinded to patients diagnosis and outcome. A third reader will solve discrepancies between the two readers. They will fill in a standardized LUS and FASH report.

AI-evaluated LUS and FASH The US images will be further used for secondary studies developing deep learning algorithms for LUS and FASH diagnosis.

Follow-up (D7 and D28) Patients will receive a follow-up phone call by the study nurse on day 7 and day 28. Data on the clinical evolution are collected: hospitalization, non-invasive ventilation, intubation, death.

Follow-up of TB treatment failures and deaths until D180 TB patients will be followed in the national TB register and treatment failures will be recorded at 6 months of treatment (according to national guidelines).

Deaths will be recorded until D180 as well.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Suspicion of lower respiratory tract infection (defined as presence of cough with at least one of the following: fever, dyspnea/tachypnea, sputum production, chest pain, hemoptysis or cachexia)

Exclusion Criteria:

* Cough/dyspnea from a definite non-infectious origin (cardiac, asthmatic...)
* Inability to cooperate with ultrasound procedure
* Inability to sign informed consent (third witness procedure available for illiterate patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Benin: 6'500 cumulative total detected and declared COVID-19 cases since march 2020 to date (NB true COVID-19 incidence unknown due to undertesting), TB incidence 55/100'000/year, low HIV (prevalence < 2%)
  * South Africa: 1,522'697 cumulative total detected and declared COVID-19 cases since march 2020 to date TB incidence 615/100.000/year, high HIV (prevalence approximately 20%)
  * Mali: 30'420 cumulative total detected and declared COVID-19 cases since march 2020 to date (NB true COVID-19 incidence unknown due to undertesting), TB incidence 52/100'000/year, low HIV (prevalence < 2%)
Sampling Method: Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity of LUS for the detection of TB | 18 to 24 months
  For LUS, each lung quadrant will be scored using a 6 feature LUS score (modified Soldati score) ranging from 1 (aerated lung), 2 (interstitial syndrome), 3 (sub centimeter pleural lesions), 4 (lung consolidation), 5 (pleural effusion) to 6 (pneumothorax). Sensitivity of LUS score for the diagnosis of TB using microbiological tests (GenXpert MTB/RIF for HIV negative patients, mycobacterial culture for HIV patients and extra-pulmonary samples) as reference standards
Specificity of LUS for the detection of TB | 18 to 24 months
  For LUS, each lung quadrant will be scored using a 6 feature LUS score (modified Soldati score) ranging from 1 (aerated lung), 2 (interstitial syndrome), 3 (sub centimeter pleural lesions), 4 (lung consolidation), 5 (pleural effusion) to 6 (pneumothorax). Sensitivity of LUS score for the diagnosis of TB using microbiological tests (GenXpert MTB/RIF for HIV negative patients, mycobacterial culture for HIV patients and extra-pulmonary samples) as reference standards
Sensitivity of FASH PLUS for the detection of TB | 24 to 36 months
  For the pericardial and abdominal ultrasound, a score according to the FASH PLUS protocol will be attributed ranging from 0 (no pathology) to 6 (presence of pericardial effusion, abdominal adenopathies, pleural effusion, splenic lesions, hepatic lesions, ascites). Sensitivity of FASH PLUS score for the diagnosis of TB using microbiological tests (GenXpert MTB/RIF for HIV negative patients, mycobacterial culture for HIV patients and extra-pulmonary samples) as reference standards.
Specificity of FASH PLUS for the detection of TB | 24 to 36 months
  For the pericardial and abdominal ultrasound, a score according to the FASH PLUS protocol will be attributed ranging from 0 (no pathology) to 6 (presence of pericardial effusion, abdominal adenopathies, pleural effusion, splenic lesions, hepatic lesions, ascites). Specificity of FASH PLUS score for the diagnosis of TB using microbiological tests (GenXpert MTB/RIF for HIV negative patients, mycobacterial culture for HIV patients and extra-pulmonary samples) as reference standards.
Sensitivity of combined LUS and FASH PLUS features for the detection of TB | 24 to 36 months
  Sensitivity of combined LUS and FASH PLUS score for the diagnosis of TB using microbiological tests (GenXpert MTB/RIF for HIV negative patients, mycobacterial culture for HIV patients and extra-pulmonary samples) as reference standards.
Specificity of combined LUS and FASH PLUS features for the detection of TB | 24 to 36 months
  Specificity of combined LUS and FASH PLUS score for the diagnosis of TB using microbiological tests (GenXpert MTB/RIF for HIV negative patients, mycobacterial culture for HIV patients and extra-pulmonary samples) as reference standards.
Sensitivity of AI-interpreted LUS for the detection of TB | 24 to 36 months
  LUS images will be scored binary by microbiological-label trained algorithms as TB or not TB. Prediction: Sensitivity of AI-assisted interpretation LUS for the detection of TB using microbiological tests as reference standards
Specificity of AI-interpreted LUS for the detection of TB | 24 to 36 months
  LUS images will be scored binary by microbiological-label trained algorithms as TB or not TB. Prediction: Specificity of AI-assisted interpretation LUS for the detection of TB using microbiological tests as reference standards
Sensitivity of AI-interpreted FASH PLUS for the detection of TB | 24 to 36 months
  FASH PLUS images will be scored binary by microbiological-label trained algorithms as TB or not TB. Prediction: Sensitivity of FASH PLUS for the detection of TB using microbiological tests as reference standards
Specificity of AI-interpreted FASH PLUS for the detection of TB | 24 to 36 months
  FASH PLUS images will be scored binary by microbiological-label trained algorithms as TB or not TB. Prediction: Specificity of FASH PLUS for the detection of TB using microbiological tests as reference standards

SECONDARY OUTCOMES:
Qualitative assessment using semi-structured interviews (based on grounded theory methods) with end users of the barriers and facilitators of the implementation of POCUS | 12 months
  Qualitative assessment using semi-structured interviews (based on grounded theory methods) with end users of the barriers and facilitators of the implementation of POCUS to assess its feasibility, sustainability and acceptability
Qualitative assessment using semi-structured interviews (based on grounded theory methods) with end users of the barriers and facilitators of the implementation of AI clinical decision support | 12 months
  Qualitative assessment using semi-structured interviews (based on grounded theory methods) with end users of the barriers and facilitators of the implementation of AI clinical decision support to assess its feasibility, sustainability and acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Anne Hartley, MD-PhD, Principal Investigator — Ecole Polytechnique Fédérale de Lausanne; Noémie Boillat Blanco, MD-PhD, Principal Investigator — University of Lausanne Hospitals; Veronique Suttels, MD, Principal Investigator — University of Lausanne Hospitals
Locations (3):
- CNHUPPC, Cotonou, Atlantic, Benin
- CHU point G, Bamako, Mali
- Wits Rural University, Acornhoek, South Africa

IPD SHARING:
Plan to Share IPD: Undecided